CLINICAL TRIAL: NCT05976061
Title: High- and Low-risk Actinic Keratosis Referrals to Secondary Care. Implementation of the General Practitioners Guidelines for Actinic Keratosis Patients.
Brief Title: High- and Low-risk Actinic Keratosis Referrals to Secondary Care
Status: Active, not recruiting | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Tergooi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-2432
Record Dates: First submitted 2023-07-20; First posted 2023-08-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Actinic Keratoses
Keywords: General Practitioners guidelines; actinic keratosis; general physician; dermatology; low-risk patients; referrals
MeSH Terms: conditions — Keratosis, Actinic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Low risk patients: Low risk actinic keratosis patients referred by the general practitioner and diagnosed as actinic keratosis by the dermatologist in 2018 and 2019.
- High risk patients: High risk actinic keratosis patients referred by the general practitioner and diagnosed as actinic keratosis by the dermatologist in 2018 and 2019.

SUMMARY:
This study evaluates the implementation of the General Practitioners guidelines 'Suspicious Skin Lesions' and investigated whether their publication and implementation has led to a reduction in the proportion of referrals of low-risk patients with actinic keratosis to secondary care, after publication of the General Practitioners guidelines and implementation activities.

DETAILED DESCRIPTION:
In the Dutch healthcare system, patients are first examined by the general practitioner who decides whether a referral to a dermatologist is indicated. Both general practitioners and dermatologists can diagnose and treat patients with actinic keratosis. Therefore, it is necessary to distinguish which patients the general practitioner should refer to a dermatologist and which patients are suitable to be treated by the general practitioner.

This retrospective data study evaluates the proportion of low risk actinic keratosis patients in 2019 en 2018.

ELIGIBILITY:
Inclusion Criteria:

* patients of 18 years and older
* referred to dermatologist for suspicion of actinic keratosis and diagnosed as actinic keratosis by the dermatologist
* treated at MaastrichtUMC+ or TergooiHospital

Exclusion Criteria:

* different diagnosis than actinic keratosis
* referred by a different specialist than the general practitioner
* referred with multiple problems
* referred for a second opinion
* if the patients was treated as different diagnosis than actinic keratosis by general practitioner

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Data from patients are collected retrospectively using the Electronic health records. Patients were selected based on the diagnosis-treatment-combination (DTC) 17 (premalignant lesion) and DTC 14 (cutaneous malignancy) that was registered from January 2018 to December 2019 by the dermatologist.
Sampling Method: Non-Probability Sample
Enrollment: 3379 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in proportion of low-risk actinic keratosis patients among all actinic keratosis patients. | 2018 compared to 2019 (2 years)
  The change in proportion of low-risk actinic keratosis patients among all actinic keratosis patients referred by the general practitioner to the dermatologist. The definition of low-risk actinic keratosis patients was based on the General Practitioners guidelines 'Suspicious skin lesions' (published in 2017). Patients were defined as low-risk when they were not immunocompromised, did not have a cutaneous malignancy in their medical history, did not have previous treatment or if they did not have extensive lesions.

CONTACTS AND LOCATIONS:
Overall Officials: Klara Mosterd, prof.dr., Principal Investigator — Maastricht UMC; Maud Jansen, dr., Principal Investigator — Maastricht UMC
Locations (1):
- Ellen Oyen, Maastricht, Netherlands

REFERENCES:
- See also: the Dutch College of General Practitioners guidelines 'Suspicious Skin lesions'. [updated 2020]. — https://richtlijnen.nhg.org/standaarden/verdachte-huidafwijkingen